CLINICAL TRIAL: NCT04078854
Title: The Impact of Sexual Health and Amputation Focused Education on Regulation of Glucose and Amputation Prevention (SAFER GAP)
Brief Title: The Impact of Sexual Health and Amputation Focused Education on Regulation of Glucose and Amputation Prevention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval expired on 3/16/2022. Study would need to be reapproved by the IRB with a new submission given the duration of expiration.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-10489
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Ulcers on Both Feet; Amputation; Traumatic, Limb; Sexual Dysfunction; Diabetic Foot Ulcer Ischemic
Keywords: Diabetic Foot; Sexual Dysfunction; Amputation
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The patients will be randomized to one of the two presentations. Both presentations are identical in educating patients how to control diabetes and the risk of future amputations in diabetes, but the experimental arm presentation will also include information regarding sexual dysfunction in diabetes.
Who Masked: Participant
Masking Description: Participants do not know that there are two types of presentations. When a potential enrollee has been identified, while still inpatient, one research associate from a group of trained residents or medical students will spend 15 to 30 minutes with the patient to enroll and give one of the two education video presentations. The patients will be randomized to one of the two presentations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot amputation, sexual health (Experimental): Group 1, Experimental arm: inpatient diabetics after initial minor foot amputation, who will be shown video on diabetes and foot amputations plus sexual health
  Interventions: Behavioral: Diabetes education
- Foot amputation, no sexual health (Active Comparator): Group 2, Control arm: inpatient diabetics after initial minor foot amputation, who will be shown video on diabetes and foot amputations, with no mention about sexual health
  Interventions: Behavioral: Diabetes education

INTERVENTIONS:
Behavioral: Diabetes education — Both presentations are identical in educating patients how to control diabetes and the risk of future amputations in diabetes, but the experimental arm presentation will also include information regarding sexual dysfunction in diabetes.
  Other Names: Sexual dysfunction in diabetes

SUMMARY:
The purpose of this study is to investigate the effect of two types of education on HbA1c level and future amputations in inpatient diabetics after initial minor foot amputation

DETAILED DESCRIPTION:
This is a single center prospective randomized study evaluating inpatient diabetics after initial minor foot amputations.

b) When a potential enrollee has been identified, while still inpatient, one research associate from a group of trained residents and medical students will spend 15-30 minutes with the patient to enroll and give one of the two education video presentations. The video presentations are the narrated versions of the slides attached to the IRB application. We will have both English and Spanish videos available. Because we are using video education, the education provided will be standardized across all patients, and there will be minimal variation in education provided despite using different research associates. The patients will be randomized to one of the two presentations. Both presentations are identical in educating patients how to control diabetes and the risk of future amputations in diabetes, but the experimental arm presentation will also include information regarding sexual dysfunction in diabetes. Each enrollee will also be asked if they are receiving structured diabetes education at the Montefiore Diabetic Center and will be encouraged to follow up to receive structured education there.

The education presentation will occur after post-operative day 1 after minor foot amputations.

Primary Outcome: HbA1c level Secondary Outcomes: LDL level, Mortality, Re-amputation (higher level or contralateral leg)

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 6.5 and above
* had minor foot amputation this hospitalization
* Age 18 years old and older
* All ethnicities
* Both genders

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes all genders are eligible
Enrollment: 21 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (HbA1c) levels | 3 months, 6 months, 1 year, 2 years
  HbA1c measures the amount of blood sugar (glucose) attached to hemoglobin

SECONDARY OUTCOMES:
Change in LDL Cholesterol levels | 3 months, 6 months, 1 year, 2 years
  LDL
Number of Deaths | 3 months, 6 months, 1 year, 2 years
  Mortality
Number of amputations of lower extremities | 3 months, 6 months, 1 year, 2 years
  Amputation
Number of re-amputations | 3 months, 6 months, 1 year, 2 years
  higher level or contralateral leg
Number of patients with mobility problems | 3 months, 6 months, 1 year, 2 years
  Number of blocks patient can walk before claudication

CONTACTS AND LOCATIONS:
Overall Officials: Issam Koleilat, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No